CLINICAL TRIAL: NCT06728839
Title: Efficacy, Safety and Tolerability of Magnesium Sulfate With Low-volume Polyethylene Glycol for Bowel Preparation Before Colonoscopy: A Multicentre, Randomized, Controlled Trial
Brief Title: Efficacy, Safety and Tolerability of Magnesium Sulfate With Low-volume Polyethylene Glycol for Colonoscopy Cleansing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: The First Affiliated Hospital of Nanchang University (Other); The First Affiliated Hospital of Zhengzhou University (Other); The Second Hospital of Hebei Medical University (Other); Daping Hospital of Army Medical University (Other); Ningjin People's Hospital (Unknown); Zibo Central Hospital (Other Government); Zhengzhou Central Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Affiliated Yueqing Hospital of Wenzhou Medical University (Other); Qianfoshan Hospital (Other); The General Hospital of Western Theater Command (Other); Jiangmen Central Hospital (Other); The First Affiliated Hospital of Henan University of Science and Technology (Other); LiuZhou People's Hospital (Other); The Fifth Affiliated Hospital of Zunyi Medical College (Other); Yan'an University Affiliated Hospital (Other); 900 Hospital of Joint Logistics Support Force of PLA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: MGSP-2024
Record Dates: First submitted 2024-12-08; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Bowel Preparation for Colonoscopy
Keywords: Magnesium sulfate; colonoscopy; bowel preparation; adenoma detection rate
MeSH Terms: interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1L PEG + 50g Magnesium sulfate (Group A) (Experimental): Take 50g magnesium sulfate and 1L polyethylene glycol for bowel preparation before colonoscopy
  Interventions: Drug: 1L PEG + 50g magnesium sulfate
- 3L PEG alone (Group B) (Active Comparator): Take 3L polyethylene glycol for bowel preparation before colonoscopy
  Interventions: Drug: 3L PEG
- 4L PEG alone (Group C) (Active Comparator): Take 4L polyethylene glycol for bowel preparation before colonoscopy
  Interventions: Drug: 4L PEG

INTERVENTIONS:
Drug: 1L PEG + 50g magnesium sulfate — Subjects in Group A will use a regimen combining magnesium sulfate and polyethylene glycol for preoperative bowel preparation and undergo colonoscopy. 1 litter of polyethylene glycol is taken at 8pm the day before the colonoscopy and 50 gram of magnesium sulfate is taken 4-6 hours before the colonoscopy, and then drink 2000 ml of water within 2 hours.
  Arms: 1L PEG + 50g Magnesium sulfate (Group A)
Drug: 3L PEG — Subjects in Group B will use a regimen with 3L polyethylene glycol for preoperative bowel preparation and undergo colonoscopy. The 3 liters of polyethylene glycol solution is taken in split dosing, with 1 liter taken at 8pm the day before the colonoscopy and 2 liters taken 4-6 hours before the colonoscopy.
  Arms: 3L PEG alone (Group B)
Drug: 4L PEG — Subjects in Group C will use a regimen with 4L polyethylene glycol for preoperative bowel preparation and undergo colonoscopy. The 4 liters of polyethylene glycol solution is taken in split dosing, with 2 liters taken at 8pm the day before the colonoscopy and 2 liters taken 4-6 hours before the colonoscopy.
  Arms: 4L PEG alone (Group C)

SUMMARY:
Magnesium salts such as magnesium citrate are often combined with polyethylene glycol to make the intestinal preparation before colonoscopy, which has shown high cleaning efficacy. Magnesium sulfate combined with polyethylene glycol is less used in the world. This multicenter, randomized, controlled trial is aimed at to evaluate the efficacy and safety of magnesium sulfate combined with low-volume polyethylene glycol for preoperative bowel preparation for colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old, male or female
* To undergo screening, surveillance and diagnostic colonoscopy
* Signed written informed consent

Exclusion Criteria:

* Subjects with therapeutic colonoscopy for colorectal polyps
* Subjects with confirmed or suspected gastrointestinal obstruction, gastric retention, gastroparesis, gastric emptying disorder, or acute gastrointestinal bleeding
* Subjects with confirmed or suspected colorectal cancer, inflammatory bowel disease, toxic colitis, or toxic megacolon
* Subjects with renal or liver dysfunction, congestive heart failure or rhabdomyolysis
* Subjects with ascites, suspected electrolyte abnormalities, or uncorrected dehydration
* Subjects with constipation (<3 times a week, difficult defecation, dry stool, less amount)
* Subjects with serious cardiac and cerebrovascular diseases,suffering from metabolic disease or endocrine disease
* Subjects who had previously undergone colorectal resection
* Women with positive pregnancy tests or pregnancy plans, and women in lactation or allergic to the investigational drugs and their ingredients
* Subjects who are participating in other clinical trials or receiving special drugs
* Subjects with any other conditions that the investigator considered inappropriate for inclusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1329 (Estimated)
Dates: Start 2024-12-09 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Adequate bowel preparation rate | 30minutes
  Defined as the proportion of participants with score ≥ 2 for all colon segment (right-side colon, transverse colon, and left-side colon) according to the Boston Bowel Preparation Scale

SECONDARY OUTCOMES:
Excellent bowel preparation rate | 30minutes
  The proportion of participants with total score ≥ 8 according to Boston Bowel Preparation Scale.
BBPS score (including total score, left colon, transverse colon, and right colon) | 30minutes
Adenoma detection rate | 10 days
Bowel preparation completion rate | 30minutes
Electrolyte levels | 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Li, MD, Principal Investigator — Changhai Hospital

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Ge F, Kang X, Wang Z, Zhu H, Liao L, Wang M, Jia J, Lou L, Guo X, Pan Y, Wan J. Low-dose of magnesium sulfate solution was not inferior to standard regime of polyethylene glycol for bowel preparation in elderly patients: a randomized, controlled study. Scand J Gastroenterol. 2023 Jan;58(1):94-100. doi: 10.1080/00365521.2022.2106154. Epub 2022 Aug 3. PMID 35920250
- [Background] Park SS, Sinn DH, Kim YH, Lim YJ, Sun Y, Lee JH, Kim JY, Chang DK, Son HJ, Rhee PL, Rhee JC, Kim JJ. Efficacy and tolerability of split-dose magnesium citrate: low-volume (2 liters) polyethylene glycol vs. single- or split-dose polyethylene glycol bowel preparation for morning colonoscopy. Am J Gastroenterol. 2010 Jun;105(6):1319-26. doi: 10.1038/ajg.2010.79. Epub 2010 May 18. PMID 20485282